CLINICAL TRIAL: NCT06207019
Title: Post-Operative Pain Evaluation After Using Different Single-file Root Canal Preparation System: A Randomized Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Abdel Moneim Ahmed Elkalashy, Elkalashy AA, Tanta University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: #R-END-1-20-5
Record Dates: First submitted 2024-01-05; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Root Canal Treatment
Keywords: Hyflex/EDM; Post-operative pain; Single-file systems; Wave One Gold; XP-endo shaper.
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyflex EDM (Active Comparator): Hyflex EDM One File (25/) with variable taper was used in continuous rotation at 500 rpm and 2.5 Ncm in a circumferential brushing action in the coronal and middle thirds, then in a pecking action for three to five cycles until the WL was reached.
  Interventions: Device: Hyflex EDM , The XP-endo Shaper, Primary WaveOne Gold
- The XP-endo Shaper (Active Comparator): The XP-endo Shaper (30/0.01) was used in rotation mode at 800 rpm and 1.0 Ncm torque. Long, gentle strokes with amplitudes of 3-4 mm were used to go down to adjusted WL in three to five cycles. After it reached the WL over the adjusted WL, it was subjected to five more up-and-down motions.
  Interventions: Device: Hyflex EDM , The XP-endo Shaper, Primary WaveOne Gold
- Primary WaveOne Gold (Active Comparator): Primary WaveOne Gold (25/07) was applied three times in a reciprocating motion; a gradual in-and-out pecking movement was utilized as directed by the manufacturer till the WL was reached.
  Interventions: Device: Hyflex EDM , The XP-endo Shaper, Primary WaveOne Gold

INTERVENTIONS:
Device: Hyflex EDM , The XP-endo Shaper, Primary WaveOne Gold — rotary single files

SUMMARY:
The goal of this clinical trial is to assess post-operative pain following root canal preparation using various single-file systems

DETAILED DESCRIPTION:
The goal of this clinical trial is to assess post-operative pain following root canal preparation using various single-file systems.Postoperative pain assessment was done by an independent evaluator with no knowledge of the group under investigation. The visual Analogue Scale (VAS) was employed. Patients could put a mark anywhere on the VAS sheet with values ranging from 0 to 100 mm [10].

* Score 0: No pain (between 0 and 4 mm) the tooth after treatment felt normal, and no discomfort was reported by the patients.
* Score 1: Recognizable, mild pain (between 5 and 44 mm), not requiring analgesics.
* Score 2: Moderate pain (between 45 and 74 mm) that is uncomfortable but bearable (when analgesics were taken, the pain was successfully reduced).
* Score 3: Severe pain (between 75 and 100 mm) painful to endure (pain was not relieved by taking analgesics).

The patients in this study were not aware of the preparation system used during treatment. Following treatment, three readings were taken at 24, 72, and 7 days. Each patient carried a VAS form, and reminder calls were made to record pain levels and return the form filled out completely

ELIGIBILITY:
Inclusion Criteria:

* • Teeth with a single root canal with nearly the same apical diameter (#15)

  * Vital pulp exposures due to caries or trauma with asymptomatic pulpitis
  * Restorable teeth

Exclusion Criteria:

* • Patients with immune deficiencies or systemic illnesses

  * Pregnant women
  * Cases of re-treatment
  * Symptomatic non-vital teeth that require root canal therapy
  * Presence of root resorption
  * Teeth with anatomic variations
  * A cute periapical abscess cases with pus discharge
  * A patient who has several teeth that need to be treated in order to eliminate the likelihood of pain referral
  * Periodontal diseases
  * Patients on analgesics, anti-inflammatory drugs, sedatives, or antibiotics seven days before therapy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain evaluation | 24 hours to 7 days
  Postoperative pain assessment was done by an independent evaluator with no knowledge of the group under investigation. The visual Analogue Scale (VAS) was employed. Patients could put a mark anywhere on the VAS sheet with values ranging from 0 to 100 mm [10]. • Score 0: No pain (between 0 and 4 mm) the tooth after treatment felt normal, and no discomfort was reported by the patients. • Score 1: Recognizable, mild pain (between 5 and 44 mm), not requiring analgesics. • Score 2: Moderate pain (between 45 and 74 mm) that is uncomfortable but bearable (when analgesics were taken, the pain was successfully reduced). • Score 3: Severe pain (between 75 and 100 mm) painful to endure (pain was not relieved by taking analgesics). The patients in this study were not aware of the preparation system used during treatment. Following treatment, three readings were taken at 24, 72, and 7 days. Each patient carried a VAS form, and reminder calls were made to record pain levels and return the form fill

CONTACTS AND LOCATIONS:
Overall Officials: Abdel Moneim A. Elkalashy, Assis.lecturer, Principal Investigator — Assis.lecturer at endodontic department
Locations (1):
- Faculty of Dentistry, Tanta University, Egypt, Tanta, Gharbia Governorate, Egypt